CLINICAL TRIAL: NCT04405271
Title: Randomized, Double-blind, Placebo-controlled Trial of TAF/FTC for Pre-exposure Prophylaxis of COVID-19 in Healthcare Workers (CoviPrep Study)
Brief Title: TAF/FTC for Pre-exposure Prophylaxis of COVID-19 in Healthcare Workers (CoviPrep Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Vaccine availability precluded further recruitment
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Sociedad Argentina de Infectología (SADI) (Argentine Society of Infectious Diseases) (Unknown)
Responsible Party: Principal Investigator, Waldo Horacio Belloso, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5616
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2020-07

CONDITIONS: Healthcare Workers; COVID-19; SARS-CoV 2
Keywords: SARS Virus, SARS-CoV-2, COVID-19, Health Personnel
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment will be the same in both arms: 1 tablet per day will be administered for a total of 12 weeks. Placebo and the active principle will be indistinguishable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FTC/TAF (Experimental): Emtricitabine/Tenofovir alafenamide (FTC/TAF) in 200 mg/25 mg tablets. A dose of 1 tablet per day will be administered for a total of 12 weeks.
  Interventions: Drug: Emtricitabine/Tenofovir Alafenamide 200 MG-25 MG Oral Tablet
- Placebo (Placebo Comparator): Identical tablets to the active experimental tablets with the same characteristics and packaging. A dose of 1 tablet per day will be administered for a total of 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emtricitabine/Tenofovir Alafenamide 200 MG-25 MG Oral Tablet — Emtricitabine/Tenofovir alafenamide (FTC/TAF) in 200 mg/25 mg tablets. A dose of 1 tablet per day will be administered for a total of 12 weeks
  Other Names: FTC/TAF
  Arms: FTC/TAF
Drug: Placebo — A dose of 1 tablet per day will be administered for a total of 12 weeks.
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
A randomized parallel double-blinded placebo-controlled clinical trial to evaluate the effect of Emtricitabine/Tenofovir alafenamide (FTC/TAF) compared with placebo on the risk of developing SARS-CoV-2 disease (COVID-19) in healthcare workers with high transmission risk in addition to currently recommended control measures.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled clinical trial. Phase III clinical trial for a new indication

Rationale One of the most affected subgroups during the current pandemic is represented by healthcare workers. In Argentina between 14 and 17% of the total COVID-19 cases are represented by this subgroup. In this sense, it appears as an adequate strategy testing the efficacy of pharmacological PrEP approaches on top of the currently recommended control measures.

The use of placebo is warranted for two main reasons: all healthcare workers will be allowed and encouraged to comply with non-pharmacological infection control measures for the protection of viral transmission. On the other hand, the use of a blinded placebo is intended for avoiding relaxation of the non-pharmacological control measures.

Tenofovir has been identified by both docking and in vitro studies as an inhibitor of RdRp (RNA dependent RNA polymerase) of coronavirus.

FTC/TAF has the additional advantage that is already being used in a pre-exposure prophylaxis setting and its safety is widely known.

Main objective To evaluate the risk of developing SARS-CoV-2 disease (COVID-19) in healthcare workers with high transmission risk in addition to currently recommended control measures.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare workers voluntarily deciding to participate in the study
2. Understanding the study purpose
3. Having between 18 and 70 years old
4. Having a high transmission risk for Covid-19. Physicians, nurses, lab technicians, physical therapists, or cleaning personnel working at COVID-19 areas, hospital emergency areas, or Intensive care units from healthcare institutions with the direct assistance of patients with Covid-19.
5. Not having a prior diagnosis of SARS-CoV-2 infection (COVID-19)
6. Having a negative IgM/IgG antibodies test for SARS-CoV-2 (COVID-19) prior to study entry
7. Negative pregnancy test for childbearing age women within 7 days prior to study entry.
8. Childbearing age males and females should comply with the use of a proven contraceptive method (double barrier methods, oral contraceptives or contraceptive hormone implants) during the course of the study and at least one month after study completion.

Exclusion Criteria:

1. Having symptoms compatible with COVID-19
2. Diagnosed HIV infection
3. Current use of Pre-exposure prophylaxis for HIV
4. Diagnosed Hepatitis B infection.
5. Diagnosed renal insufficiency and or current hemodialysis need
6. Diagnosed osteoporosis under pharmacological treatment.
7. Weight < 40kg
8. Current immunosuppressive or serious hematological condition
9. Prior use of pre-exposure prophylaxis for SARS-CoV-2
10. Current pregnancy or pregnancy plan within the study course.
11. Current breastfeeding
12. Known hypersensitivity to any of the study medication components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1378 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
COVID-19 incident cases | During treatment (12 weeks)
  SARS-CoV-2 disease (COVID-19) with or without symptoms at week 12 of treatment as defined by the presence of specific antibodies against the virus. Positive cases will be confirmed by PCR

SECONDARY OUTCOMES:
Number of asymptomatic SARS-CoV-2 (Covid-19) infections confirmed by serology | During treatment (12 weeks)
  Number of asymptomatic SARS-CoV-2 (Covid-19) infections confirmed by serology
Severity of symptomatic COVID-19 | During treatment (12 weeks)
  Severity of symptomatic SARS-CoV-2 (Covid-19) infections as defined by the following categories:
  * Mild symptoms: malaise, fever, cough, arthralgia myalgias,
  * Moderate symptoms: same as above plus shortness of breath
  * Severe symptoms: clinical status requiring admission in Intensive care unit
Respiratory symptom duration in days | During treatment (12 weeks)
  Respiratory symptom duration in days
Relation between treatments and symptoms duration | During treatment (12 weeks)
  Relation between treatments and symptoms duration
Time course of specific IgM/IgG seroconversion | During treatment (12 weeks)
  Time course of specific IgM/IgG seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: Waldo H Belloso, MD, Study Chair — Hospital Italiano de Buenos Aires; Ventura Simonovich, MD, Principal Investigator — HIBA; Esteban Nannini, MD, Principal Investigator — Sanatorio Britanico; Wanda Cornistein, MD, Principal Investigator — Hospital Austral; Marcelo Figueiras, MD, Principal Investigator — Richmond Laboratorio; Elvira Zini, MD, Principal Investigator — Richmond Laboratorio; Fernando Riera, MD, Principal Investigator — Sanatorio Allende (Córdoba); Omar Sued, MD, Principal Investigator — HUESPED; Santiago Ramirez Borga, MD, Principal Investigator — Hospital Italiano de La Plata; Gustavo Costilla Campero, MD, Principal Investigator — Hospital Padilla (Tucumán); Gustavo D Lopardo, MD, Principal Investigator — Hospital Bernardo Houssay; Gonzalo Corral, MD, Principal Investigator — Hospital Alende (Mar del Plata)
Locations (1):
- Sociedad Argentina de Infectología, A. J. Carranza 974, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elfiky AA. Anti-HCV, nucleotide inhibitors, repurposing against COVID-19. Life Sci. 2020 May 1;248:117477. doi: 10.1016/j.lfs.2020.117477. Epub 2020 Feb 28. PMID 32119961
- [Background] Castillo-Mancilla JR, Meditz A, Wilson C, Zheng JH, Palmer BE, Lee EJ, Gardner EM, Seifert S, Kerr B, Bushman LR, MaWhinney S, Anderson PL. Reduced immune activation during tenofovir-emtricitabine therapy in HIV-negative individuals. J Acquir Immune Defic Syndr. 2015 Apr 15;68(5):495-501. doi: 10.1097/QAI.0000000000000529. PMID 25763783
- See also: Sala de Situación Coronavirus online - Ministerio de Salud de la Nación — https://www.argentina.gob.ar/salud/coronavirus-COVID-19/sala-situacion
- See also: Reasons for healthcare workers becoming infected with novel coronavirus disease 2019 (COVID-19) in China — https://doi.org/10.1016/j.jhin.2020.03.002
- See also: Nucleotide Analogues as Inhibitors of SARS-CoV-2 Polymerase — https://doi.org/10.1101/2020.03.18.997585
- See also: Nucleotide Analogues as Inhibitors of Viral Polymerases — https://www.biorxiv.org/content/biorxiv/early/2020/01/31/2020.01.30.927574.full.pdf
- See also: Triphosphates of the Two Components in DESCOVY and TRUVADA are Inhibitors of the SARS-CoV-2 Polymerase — https://doi.org/10.1101/2020.04.03.022939
- See also: THE PHASE 3 DISCOVER STUDY: DAILY F/TAF OR F/TDF FOR HIV PREEXPOSURE PROPHYLAXIS — https://www.croiconference.org/abstract/phase-3-discover-study-daily-ftaf-or-ftdf-hiv-preexposure-prophylaxis/
- See also: 1962. Renal Outcomes for Participants Taking F/TAF vs. F/TDF for HIV PrEP in the DISCOVER Trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6808931/